CLINICAL TRIAL: NCT00956397
Title: Does Small Intestinal Bacterial Overgrowth Contribute to Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry C. Lin, MD (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Henry C. Lin, MD, Henry C. Lin, MD, New Mexico VA Healthcare System
Organization: New Mexico VA Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRRC 07-187; 5R21DK078101-02 (NIH)
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Functional Dyspepsia; Small Intestinal Bacterial Overgrowth; Chronic Abdominal Discomfort
Keywords: Functional Dyspepsia; Small Intestinal Bacterial Overgrowth; chronic abdominal discomfort
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Participants (Active Comparator)
  Interventions: Procedure: Lactulose Breath Test
- FD Participants (Active Comparator)
  Interventions: Drug: Rifaximin; Procedure: Lactulose Breath Test
- FD (Placebo) Participants (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — rifaximin 550 mg TID PO x 10 days
  Other Names: Xifaxan
  Arms: FD Participants
Procedure: Lactulose Breath Test — Test will begin with a baseline breath sample followed by ingestion of 10g of lactulose (Xactdose, South Beloit, IL) in 100ml of water. Breath samples will be collected every 15 min for 180 min. Gas samples will be analyzed for hydrogen and methane using a gas chromatograph (Model SC, Quintron Instruments, Milwaukee, WI).
  Arms: Control Participants; FD Participants
Drug: Placebo — placebo TID x 10 days
  Arms: FD (Placebo) Participants

SUMMARY:
The prevalence of functional dyspepsia (FD) is estimated to be 15% of the adult population. FD is commonly described as a condition of chronic abdominal discomfort localized to the upper abdomen. Postprandial bloating, pain, nausea, vomiting, belching, and early satiety are common symptoms of the FD patient. FD is defined by >12 weeks of symptoms, which need not be consecutive, within the preceding year consisting of a) persistent or recurrent dyspepsia and b) an absence of organic disease after a gastrointestinal endoscopy or x-ray series. FD is therefore considered a disorder of function because no mucosal pathology is seen in these patients, as in patients with other functional disorders such as irritable bowel syndrome (IBS) and fibromyalgia (FM). There is a remarkable degree of overlap among these three disorders. These 3 disorders share the finding of hypersensitivity and the symptom of postprandial bloating to suggest the possibility of a common origin.

ELIGIBILITY:
Inclusion Criteria:

* Must have FD based on the most recent Umbrella criteria of one or more of: a. bothersome postprandial fullness, b. early satiation, c. epigastric pain, d. epigastric burning
* No evidence of organic disease (including H. pylori detected at time of endoscopy) that is likely to explain the symptoms
* Criteria must be fulfilled for the last 3 months with symptom onset at least 6 months before the diagnosis
* The physical exam, routine blood tests including CBC, chemistry panel and liver tests, upper gastrointestinal endoscopy and 24h pH study must be normal

Exclusion Criteria:

* History of IBS,rheumatoid arthritis,H. Pylori infection,lupus,peptic ulcer, cirrhosis,diabetes, HIV or TB
* Inflammatory bowel disease
* Bowel Resection (including gastric, small bowel or colon; gallbladder surgery or appendectomy are NOT exclusion criteria)
* Anti/pro-biotics last 3 months
* Previous LBT (Lactulose Breath Test)
* Narcotic Dependence
* Pregnancy
* Control subjects will be excluded if they have symptoms of heartburn, retrosternal chest pain, chronic cough, nausea or regurgitation suggestive of gastroesophageal reflux disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To compare the pattern of bacterial gas excretion in breath among Veterans with FD vs. controls using LBT | every 15 minutes for 180 minutes

SECONDARY OUTCOMES:
The investigators will determine the relationship between SIBO in FD patients using randomized antibiotic treatment | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henry C Lin, MD, Principal Investigator — New Mexico VA Healthcare System
Locations (1):
- General Clinical Research Center, Albuquerque, New Mexico, United States